CLINICAL TRIAL: NCT00227383
Title: Effect of Electroacupuncture in Diabetic Patients With Gastroparesis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Medical University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DMR94-IRB-69
Record Dates: First submitted 2005-09-27; First posted 2005-09-28 (Estimated); Last update posted 2007-01-22 (Estimated); Status verified 2005-09

CONDITIONS: Diabetes Mellitus; Gastroparesis
Keywords: Diabetes; gastroparesis; electroacupuncture
MeSH Terms: conditions — Diabetes Mellitus; Gastroparesis | interventions — Electroacupuncture

INTERVENTIONS:
Device: Electroacupuncture (device)

SUMMARY:
In this study, we aim at evaluating the effect of electroacupuncture in diabetic patients with gastroparesis. Patient-based symptom severity measure, serum parameters and solid-phase gastric emptying time are measured to evaluate the effectiveness of electroacupuncture.

DETAILED DESCRIPTION:
Initially, we will collect 30 patients with type 2 diabetes with a ≧ 3-month history of dyspeptic symptoms. An upper GI endocopy will be obtained to rule out possibility of organic obstruction. Cardiac arrhythmia and pregnancy will be excluded. None of them ever received abdominal surgery. Patients are then randomized to one of two treatment arms. Arm I: 15 patients received EA stimulation on acupoints St-36 (Zusanli) and Li-4 (Hegu). Arm II: 15 subjected to EA stimulation on non-acupoints around St-36 and Li-4 with the same electrical pulse and amplitude. Gastroparesis Cardinal Symptom Index (GCSI) and solid-phase gastric emptying time will be measured on baseline and after EA. In addition, serum gastrin, motilin, human pancreatic polypeptide, fasting blood sugar, and postprandial glucose levels will be also monitored.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Dyspetic symptoms for more than 3 months
* Symptoms include nausea, vomiting, upper abdominal discomfort, early satiety, bloating and anorexia

Exclusion Criteria:

* Organic gastrointestinal obstruction
* Previous surgery of gastrointestinal tract
* Cardiac arrhythmia
* Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30

PRIMARY OUTCOMES:
Solid-phase gastric emptying time and score on Gastroparesis Cardinal Symptom Index(GCSI) at 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Pang Wang, MD, Study Chair — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan